CLINICAL TRIAL: NCT03808337
Title: PROMISE-005: A Phase II Randomized Study Assessing the Efficacy of Stereotactic Body Radiotherapy (SBRT) in Patients With Oligometastatic Breast or Lung Cancer
Brief Title: Investigating the Effectiveness of Stereotactic Body Radiotherapy (SBRT) in Addition to Standard of Care Treatment for Cancer That Has Spread Beyond the Original Site of Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-486
Record Dates: First submitted 2019-01-16; First posted 2019-01-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer; Non Small Cell Lung Cancer; Metastatic Breast Cancer; Metastatic Non-Small Cell Lung Carcinoma
Keywords: Stereotactic body radiotherapy; SBRT; 18-486; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standare of Care (Active Comparator): Patients with newly diagnosed metastatic non-small cell lung cancer or triple negative breast cancer may be enrolled on protocol prior to receiving any systemic therapy. If these patients are randomized to the standard of care arm (Arm 1), they will initiate appropriate therapy as determined by their oncologist. Standard of care systemic therapy, including chemotherapeutics, targeted therapies, immunomodulatory agents, and hormonal therapies will be delivered at the discretion of the treating oncologist.
  Interventions: Drug: Systemic Therapy/Standard of Care
- Stereotactic Body Radiotherapy (SBRT) + Standard of Care (Experimental): Patients enrolled on Arm 2 of the study will undergo Stereotactic Body Radiotherapy/SBRT to all known metastases seen on imaging studies performed prior to enrollment. Radiotherapy will be given concurrently to all metastatic sites. Minimum BED for ablative SBRT is more than or equal to 48 Gy10. Patients can undergo systemic therapy concurrently with SBRT at the discretion of treating radiation oncologist and medical oncologist. After completion of SBRT to all sites of known metastatic disease, patients will continue standard of care therapy per the treating oncologist.
  Interventions: Radiation: Stereotactic Body Radiotherapy/SBRT; Drug: Systemic Therapy/Standard of Care

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy/SBRT — Radiation to each metastatic site should be delivered to a minimum dose of 30 Gy in 5 fractions (BED of 48 Gy10). The exact dose of radiotherapy will be determined by the treating radiation oncologist. Preferred regimens for lung metastases include 50 Gy in five fractions, 48 Gy in four fractions, or 54 Gy in three fractions, although lower doses may be employed to respect dose limits to critical structures such as the esophagus. Recommended SBRT dosing for other sites includes 27 to 30 Gy in three fractions or 24 Gy in one fraction for bone metastases.
  Arms: Stereotactic Body Radiotherapy (SBRT) + Standard of Care
Drug: Systemic Therapy/Standard of Care — Standard of care systemic therapy, including chemotherapeutics, targeted therapies, immunomodulatory agents, and hormonal therapies will be delivered at the discretion of the treating oncologist. For patients randomized to receive SBRT, systemic therapy can be continued during SBRT at the discretion and concensus of treating physicians (medical oncologist and radiation oncologist). If the treating physicians recommend discontinuing systemic therapy during SBRT, general guidelines for stopping and reinitiating systemic regimen are as follows: Hormonal therapies and immunotherapy can be continued during SBRT. Consideration can be given to holding cytotoxic chemotherapy beginning 3 to 7 days prior to the initiation of SBRT until 3 to 7 days after the completion of SBRT. Similarly, consideration can be given to holding biologic agents during SBRT and for 0 to 3 days before and after.

SUMMARY:
This study is being done to determine if stereotactic body radiotherapy (SBRT) when delivered to all sites of disease in participants with 1-5 metastases will increase the length of time before participants' disease gets worse.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic disease detected on imaging and histologically confirmed

  * Metastatic breast cancer (all subtypes)
  * Non-small cell lung cancer (NSCLC) without known targetable molecular alterations in EGFR, ALK, or ROS1
  * NSCLC with EGFR, ALK, or ROS1 targetable molecular alterations who had a history of disease progression on first-line tyrosine kinase inhibitor
* Patient can either have newly diagnosed metastatic disease, or have non-progressive disease on systemic therapy (for at least 3 months on systemic imaging)
* Patients must have measurable disease at baseline (RECIST or PERCIST 2.0) and with 5 or fewer discrete disease sites that are technically amendable to SBRT (with the exception that if the primary disease is not amendable to SBRT it is allowed to be treated with conventionally fractionated or hypfractionated radiotherapy).

  * Two lesions in such close proximity to one another that treatment with one isocenter is more accurate and safer in the liver, lungs, or other similar anatomic locations should be viewed as one site of metastatic disease treatment
  * Disease in 2 contiguous vertebral bodies (with up to 6 cm of paraspinal extension) can represent one site of disease in the spine; non-contiguous lesions in vertebral bodies separated by one vertebral body free of disease should be viewed as 2 sites of treatment
  * If the clinical scenario deem that other forms of local therapy may be more suitable for the metastatic disease, such as surgical resection and interventional radiology-guided ablation, patients would be able to undergo other forms of local therapy with discussion with the PI.
* For de novo stage IV patients (patients with metastatic disease at first presentation), primary disease must be treatable with local therapy. If the primary tumor or other locoregional disease has not been definitively treated and is not amendable to SBRT, it must be treated with conventionally fractionated or hypofractionated radiotherapy using a regimen that delivers a minimum BED of 48 Gy10. If the clinical scenario deem that other forms of local therapy may be more suitable for the primary and locoregional disease, such as surgical resection and interventional radiology-guided ablation, patients would be able to undergo other forms of local therapy with discussion with the PI.
* If primary disease was previously treated with local therapy in the form of surgery or radiation, any new local/regional disease recurrence should be technically treatable with SBRT or hypofractionated radiation. If the clinical scenario deem that other forms of local therapy may be more suitable for the local/regional recurrent disease, such as surgical resection and interventional radiology-guided ablation, patients would be able to undergo other forms of local therapy with discussion with the PI.
* Patients may receive palliative radiotherapy for symptomatic metastases or primary disease prior to enrollment provided that there is at least one other non-irradiated lesion amenable to SBRT at the time of enrollment.
* Patients with brain metastases are eligible if these lesions have been treated prior to enrollment.
* ECOG Performance status 0 - 2.
* Age >/= 18 years.
* Able to provide informed consent.
* Female subjects must either be of non-reproductive potential (i.e. post-menopausal by history: >/= 60 years old or no menses for 1> year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test within 2 weeks prior to starting treatment.
* Adequate baseline organ function to allow SBRT to all relevant targets, as determined by the treating radiation oncologist based on lesion location, lesion size, and proximity to relevant organs at risk.

Exclusion Criteria:

* Serious medical co-morbidities precluding radiotherapy, determined at the discretion of the treating investigator.
* Pregnant or lactating women.
* Other active malignancy within the last year, even if without evidence of disease.
* Clinical or radiological evidence of spinal cord compression
* Malignant pleural effusion or ascites.
* Patients whose entry to the trial will cause unacceptable clinical delays in their planned management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Up to 2 years
  To determine whether stereotactic body radiotherapy to all sites of metastatic disease in patients with oligometastatic non-small cell lung cancer or triple-negative breast cancer improves progression free survival (PFS), defined as time from randomization to disease progression or death, as compared to standard of care therapy alone.

SECONDARY OUTCOMES:
Overall Survival | Up to 2 years
  To compare overall survival (OS) between standard of care and SBRT arms.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Xu, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - Natera, Inc. (Data and Specimen Analysis Only), San Carlos, California
  - Hartford Healthcare, Hartford, Connecticut
  - WCHN Norwalk Hospital - Data Collection, Norwalk, Connecticut
  - Baptist Alliance - McI, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org